CLINICAL TRIAL: NCT01505569
Title: Alkylator-Intense Conditioning Followed by Autologous Transplantation for Patients With High Risk or Relapsed Solid or CNS Tumors
Brief Title: Auto Transplant for High Risk or Relapsed Solid or CNS Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011OC057; MT2011-09C (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Ewing's Family Tumors; Renal Tumors; Hepatoblastoma; Rhabdomyosarcoma; Soft Tissue Sarcoma; Primary Malignant Brain Neoplasms; Retinoblastoma; Medulloblastoma; Supra-tentorial Primative Neuro-Ectodermal Tumor (PNET); Atypical Teratoid/Rhabdoid Tumor (AT/RT); CNS Tumors; Germ Cell Tumors
Keywords: autologous transplantation; high risk solid tumor; relapsed solid tumor
MeSH Terms: conditions — Carcinoma, Renal Cell; Hepatoblastoma; Rhabdomyosarcoma; Sarcoma; Brain Neoplasms; Retinoblastoma; Medulloblastoma; Rhabdoid Tumor; Central Nervous System Neoplasms; Neoplasms, Germ Cell and Embryonal | interventions — Ifosfamide; Etoposide; etoposide phosphate; Mesna; Granulocyte Colony-Stimulating Factor; Busulfan; Melphalan; Thiotepa; Radiation; Carboplatin; Paclitaxel; Leukapheresis; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm A: Patients with High Risk or Relapsed Solid Tumor (Other): Treatment consists of a mobilization chemotherapy (ifosfamide 1.8 g/m^2/day intravenously [IV], etoposide 100 mg/mg^2 IV, mesna 1.8 g/m^2 divided in every 6 hours dosing, and granulocyte colony stimulating factor 10 mcg/kg subcutaneously or IV until absolute neutrophils > 1,000/mm^2) for 5 days in a 30-100 day pretransplant window, busulfan (1.1 mg/kg IV every 6 hours on days -8 through -6), melphalan (50 mg/mg^2 on days -5 and -4), thiotepa conditioning (250 mg/m^2 IV over 2 hours on days -3 and -2) followed by an autologous peripheral blood stem cell transplant (infusion on Day 0) and, if appropriate, disease specific radiation therapy at day +60.
  Interventions: Drug: Ifosfamide; Drug: Etoposide; Drug: Mesna; Biological: G-CSF; Drug: Busulfan; Drug: Melphalan; Drug: Thiotepa; Biological: Autologous stem cell infusion; Radiation: Radiation
- Arm B: Certain CNS Tumors (Other): Treatment consists of a mobilization chemotherapy (ifosfamide 1.8 g/m^2/day intravenously [IV], etoposide 100 mg/mg^2 IV, mesna 1.8 g/m^2 divided in every 6 hours dosing, and granulocyte colony stimulating factor 10 mcg/kg subcutaneously or IV until absolute neutrophils > 1,000/mm^2) for 5 days in a 30-100 day pretransplant window, carboplatin (dose based on GFR and age 17 mg/kg/day IV or 510 mg/m^2/day IV) , thiotepa conditioning (10 mg/kg/day or 300 mg/m^2 IV on days -3 and -2) followed by an autologous peripheral blood stem cell transplant (infusion on Day 0). This will be repeated up to 2 additional 30 day cycles.
  Interventions: Drug: Ifosfamide; Drug: Etoposide; Drug: Mesna; Biological: G-CSF; Drug: Thiotepa; Biological: Autologous stem cell infusion; Drug: Carboplatin
- Arm C: Germ Cell Tumors (Other): 1. High-Dose Chemotherapy (3 cycles)
     * Carboplatin AUC=8 & Etoposide 400 mg/m^2 daily, days -4, -3, and -2 every 21 days
  2. Autologous Stem Cell Infusion ≥ 3 x 106 CD34+ cells/kg Day 0 Cycles 1, 2 and 3
  3. TI Chemotherapy & PBSC Collection.
     * Paclitaxel 200mg/m^2 IV over 3 hours on Day 1 every 14 days for 2 cycles
     * Ifosfamide 2000 mg/m^2 IV daily on Days 1-3 every 14 days for 2 cycles
     * Mesna 2000 mg/m^2 on Days 1-3 every 14 days for 2 cycles
     * G-CSF 10 μg/kg sub q daily on day 3 until adequate CD34+ cell collection or day 15, whichever occurs first
     * Leukapheresis starting on approx. day 11 and continued daily until reaching the collection goal of ≥ 8 x 106 CD34+ cells/kg) or day 15, whichever occurs first
  Interventions: Drug: Ifosfamide; Drug: Etoposide; Drug: Mesna; Biological: G-CSF; Biological: Autologous stem cell infusion; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Leukapheresis
- Arm D: Certain CNS Tumors (Other): 1. Mobilization Chemotherapy and PBSC Collection (day -100 to day -30)
  2. Pre-Transplant Conditioning Chemotherapy (3 cycles)
     * Day -8, -7, -6: Carboplatin as calculated from AUC of 7 approx.
     * Day -5, -4, -3: Thiotepa 10 mg/kg, Etoposide 8.3 mg/kg
     * Day 0: Autologous Hematopoietic Cell Reinfusion
     * Day +1: Begin G-CSF(filgrastim) 5 mcg/kg
  Interventions: Drug: Etoposide; Biological: G-CSF; Drug: Thiotepa; Biological: Autologous stem cell infusion; Drug: Carboplatin
- Arm E: Neuroblastoma (Other): 1. Mobilization Chemotherapy and PBSC Collection (day -100 to day -30)
  2. Pre-Transplant Conditioning Chemotherapy (day -7 to day -0)
     * Day -7: anti-seizure prophylaxis with lorazepam or levetiracetam
     * Day -6 - -3: Busulfan IV q24 hours x 4 doses
     * Day -1: Melphalan 140 mg/m2 IV
     * Day 0: Autologous Hematopoietic Cell Reinfusion
  Interventions: Biological: G-CSF; Drug: Busulfan; Drug: Melphalan; Biological: Autologous stem cell infusion; Drug: Anti-seizure prophylaxis; Drug: Ursodiol

INTERVENTIONS:
Drug: Ifosfamide — * Arms A&B: 1.8 g/m^2/day intravenously (IV) over 1 hour; given in a window of 30-100 days before transplant for 5 days before conditioning regimen
  * Arm C: 2000 mg/m^2 IV daily on Days 1-3 every 14 days for 2 cycles
  Other Names: Mitoxana; Ifex
  Arms: Arm A: Patients with High Risk or Relapsed Solid Tumor; Arm B: Certain CNS Tumors; Arm C: Germ Cell Tumors
Drug: Etoposide — * Arms A&B: 100 mg/m^2/day intravenously (IV) over 1 hour; given in a window of 30-100 days before transplant for 5 days prior to conditioning regimen.
  * Arm C: 400 mg/m^2 daily on days -4, -3, and -2 every 21 days
  * Arm D: Etoposide 8.3 mg/kg (or 250mg/m² if age >36 mos.) approx. hour 75 on days -5, -4, and -3
  Other Names: Eposin; Etopophos; Vepesid; VP-16
  Arms: Arm A: Patients with High Risk or Relapsed Solid Tumor; Arm B: Certain CNS Tumors; Arm C: Germ Cell Tumors; Arm D: Certain CNS Tumors
Drug: Mesna — * Arms A&B: 1.8 g/m^2/day divided in every 6 hrs dosing; given in a window of 30-100 days before transplant for 5 days prior to conditioning regimen.
  * Arm C: 2000 mg/m^2 IV daily on Days 1-3 every 14 days for 2 cycles
  Other Names: Uromitexan; Mesnex
  Arms: Arm A: Patients with High Risk or Relapsed Solid Tumor; Arm B: Certain CNS Tumors; Arm C: Germ Cell Tumors
Biological: G-CSF — * Arms A&B: Beginning 24 hours after treatment with ifosfamide, etoposide and mesna, administer 10 mcg/kg/day subcutaneously (SQ) or intravenously (IV) until absolute neutrophil count (ANC) is greater than (>) 1,000/mm^2. Starting that day, increase dose to 15 mcg/kg/day SQ or IV given as a single injection for 3 doses. G-CSF, 5 ug/kg/day IV as a bolus injection each evening beginning on day 0 until the ANC is >2500 x 10^9/L for 2 consecutive days. G-CSF will subsequently be restarted at 5 ug/kg/day SC or IV if the ANC falls below 1000/mm^3
  * Arm C: 10 μg/kg SQ daily beginning 6 hours after ifosfamide on day 3 until adequate CD34+ cell collection or day 15, whichever occurs first.
  * Arm D: Beginning day +1 following hematopoietic cell reinfusion, patients receive filgrastim at a dose of 5mcg/kg SQ once daily (or 5mcg/Kg IV either daily or twice daily, per institutional preference)
  * Arm E: 5 micrograms/kg/dose beginning on Day 0 and continue per institutional preference
  Other Names: Granulocyte colony-stimulating factor
Drug: Busulfan — Arm A: 1.1 mg/kg IV every 6 hours on days -8 through -6 Arm E: first dose of busulfan is dosed by mg/kg as appropriate for age and weight. Once the results of pharmacokinetic (PK) studies are known, subsequent daily doses are based upon those results,
  Other Names: Busulfex
  Arms: Arm A: Patients with High Risk or Relapsed Solid Tumor; Arm E: Neuroblastoma
Drug: Melphalan — Arm A: 50 mg/m^2 intravenously (IV) over 30 min on Days -4 and -5 Arm E:140 mg/m2 AT LEAST 24 hrs after last busulfan dose. Day: -1
  Other Names: 50 mg/m2 IV over 30 min
  Arms: Arm A: Patients with High Risk or Relapsed Solid Tumor; Arm E: Neuroblastoma
Drug: Thiotepa — Arm A: 250 mg/m^2 intravenously (IV) over 2 hrs on days -2 and -3 Arm B: 10 mg/kg/day or 300 mg/m^2 IV on days -3 and -2 Arm D: Thiotepa 10 mg/kg (or 300mg/m² if age >36 mos.) approx. hour 72 on days -5, -4, and -3
  Other Names: Thioplex
  Arms: Arm A: Patients with High Risk or Relapsed Solid Tumor; Arm B: Certain CNS Tumors; Arm D: Certain CNS Tumors
Biological: Autologous stem cell infusion — Arms A, B & C: On Day 0, stem cells will be infused immediately after thawing over 15-60 minutes per institutional guidelines.
  Arm D: On day 0, peripheral blood hematopoietic progenitor cells (PHPCs) or bone marrow cells will be thawed and re-infused about 72 hours following completion of the last dose of chemotherapy.
  Arm E: stem cells will be infused on Day 0 of Consolidation. Where the DMSO volume in the stem cell product would exceed accepted level for infusion within a 24 hour period, stem cell products may be infused over 2 days to meet this standard.
Radiation: Radiation — Arm A: If a patient is considered for post-transplant irradiation, a disease appropriate full tumor restaging should be done prior to starting.
  Whole lung irradiation (1500cGy in 10 fractions) may be given in patients with prior lung metastasis. Areas of known metastatic disease or PET areas may receive "spot" irradiation using a dose and method determined to be tolerable by radiation oncology staff. Additional radiation will be given if primary disease has not been irradiated to maximum tolerated dose.
  Arms: Arm A: Patients with High Risk or Relapsed Solid Tumor
Drug: Carboplatin — Arm B: depending on age and GFR 17mg/kg/day IV over 4 hours or 510 mg/m^2/day IV over 4 hours Arm C: AUC=8 daily on days -4, -3, and -2 every 21 days Arm D: as calculated from AUC of 7 approx. hour 0 on days -8, -7, and -6
  Other Names: Paraplatin
  Arms: Arm B: Certain CNS Tumors; Arm C: Germ Cell Tumors; Arm D: Certain CNS Tumors
Drug: Paclitaxel — Arm C: 200 mg/m2 IV over 3 hours on Day 1 every 14 days for 2 cycles
  Other Names: Taxol; Onxal
  Arms: Arm C: Germ Cell Tumors
Procedure: Leukapheresis — Arm C: Blood will be taken by a needle placed in one arm and processed through a machine, which spins the blood so that the white blood cells will be separated out in the machine for purposes of this research and the rest of the blood will be returned through a needle in the other arm.
  Arms: Arm C: Germ Cell Tumors
Drug: Anti-seizure prophylaxis — Arm E: Lorazepam OR Levetaracetam
  * Lorazepam should be given 0.02-0.05 mg/kg/dose, given 30 minutes prior to each busulfan dose and then continuing every 6 hours, maximum dose: 2 mg.
  * Levetiracetam should be given 10 mg/kg/dose PO, administered BID, staring 12 hours prior to busulfan, maximum single dose: 1000mg.
  Arms: Arm E: Neuroblastoma
Drug: Ursodiol — Arm E: 150 mg/m2/dose PO, administered BID, beginning on Day -7 and continuing a minimum of 28 days post-transplant, or until the end of Consolidation.
  Arms: Arm E: Neuroblastoma

SUMMARY:
This is a standard of care treatment guideline for high risk or relapsed solid tumors or CNS tumors consisting of a busulfan, melphalan, thiotepa conditioning (for solid tumors) or carboplatin and thiotepa conditioning (for CNS tumors) followed by an autologous peripheral blood stem cell transplant. For solid tumors, if appropriate, disease specific radiation therapy at day +60. For CNS tumors, the conditioning regimen and autologous peripheral blood stem cell transplant will be given for 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

All patients must have histological verification of malignancy at original diagnosis.

* Eligible Diseases

  * Arm A: Solid Tumor

    * Ewing's Family Tumors (ES/PNET/DSRCT) - metastatic at time of diagnosis and/or relapsed after therapy
    * Renal Tumors - relapsed (all histology - Wilm's tumor) or at diagnosis (clear cell sarcoma and Rhabdoid tumor)
    * Hepatoblastoma - metastatic at time of diagnosis and/or relapsed after therapy
    * Rhabdomyosarcoma - metastatic at time of diagnosis and/or relapsed after therapy
    * Soft Tissue Sarcoma - chemotherapy responsive metastatic disease or chemotherapy responsive relapsed disease
    * Primary Malignant Brain Neoplasms <18 years of age - at diagnosis and/or relapse
    * Retinoblastoma - disseminated at diagnosis and/or relapsed
    * CNS Lymphoma - primary or secondary CNS lymphoma.
    * Other High Risk Metastatic or Relapsed Solid Tumors - to be approved by 2 or more pediatric hematology/oncology and bone marrow transplant (BMT) physicians
  * Arm B: Certain CNS tumors

    * Medulloblastoma: Children less than 36 months (3 years) of age at time of definitive surgery (for histopathologic diagnosis) who have high risk Medulloblastoma, defined as any one of the following:

      1. > 1.5 cm2 residual disease following resection for any Medulloblastoma histology
      2. lumbar CSF cytology positive for tumor cells by analysis of fluid collected either before definitive surgery or at least 10 days after definitive surgery
      3. MRI evidence of (a) gross nodular seeding in the intracranial subarachnoid space or ventricular system distant from primary tumor site, M2; or (b) gross nodular seeding in the spinal subarachnoid space +/- evidence of intracranial seeding, M3; or (c) extraneural metastases, M4,
    * Anaplastic Histologic Variant Medulloblastoma: less than 70 years of age, any metastatic stage, with total or sub-total resection.
    * Infant Medulloblastoma: Children less than 8 months of age at the time of definitive surgery (for histopathologic diagnosis), any histology, any metastatic state, with total or sub-total resection.
    * Supra-tentorial Primative Neuro-Ectodermal Tumor (PNET): Children less than 36 months (3 years) of age at time of definitive surgery (for histopathologic diagnosis) with or without metastatic disease
    * Atypical Teratoid/Rhabdoid Tumor (AT/RT): less than 70 years of age with CNS AT/RT (with or without metastatic disease).
    * Other High Risk CNS Tumors - to be approved by 2 or more physicians (at least one oncologist and one BMT physician).
  * Arm C: Germ Cell Tumors

    * Confirmation of germ cell tumor (GCT) histology (both seminoma and nonseminoma). Tumor may have originated in any primary site. NOTE: In rare circumstances, patients will be allowed to enroll even if a pathologic diagnosis may not have been established. This would require a clinical situation consistent with the diagnosis of GCT (testicular, peritoneal, retroperitoneal or mediastinal mass, elevated tumor marker levels {HCG ≥ 500; AFP ≥ 500} and typical pattern of metastases).

      1. One or more unfavorable prognostic features for achieving a CR with conventional-dose chemotherapy. Unfavorable prognostic features include:
      2. extragonadal primary site
      3. PD following an incomplete response (IR) to first-line therapy,
      4. PD after a conventional-dose salvage (cisplatin + ifosfamide -based) regimen
  * Arm D: Certain CNS Tumor patients who can only undergo one transplant

    * Medulloblastoma: Children less than 36 months (3 years) of age at time of definitive surgery (for histopathologic diagnosis) who have high risk Medulloblastoma, defined as any one of the following:

      * > 1.5 cm2 residual disease following resection for any Medulloblastoma histology
      * lumbar CSF cytology positive for tumor cells by analysis of fluid collected either before definitive surgery or at least 10 days after definitive surgery
      * MRI evidence of (a) gross nodular seeding in the intracranial subarachnoid space or ventricular system distant from primary tumor site, M2; or (b) gross nodular seeding in the spinal subarachnoid space +/- evidence of intracranial seeding, M3; or (c) extraneural metastases, M4,
    * Anaplastic Histologic Variant Medulloblastoma: less than 70 years of age, any metastatic stage, with total or sub-total resection.
    * Infant Medulloblastoma: Children less than 8 months of age at the time of definitive surgery (for histopathologic diagnosis), any histology, any metastatic state, with total or sub-total resection.
    * Supra-tentorial Primative Neuro-Ectodermal Tumor (PNET): Children less than 36 months (3 years) of age at time of definitive surgery (for histopathologic diagnosis) with or without metastatic disease
    * Atypical Teratoid/Rhabdoid Tumor (AT/RT): less than 70 years of age with CNS AT/RT (with or without metastatic disease).
    * Other High Risk CNS Tumors including choroid plexus carcinoma in children- to be approved by 2 or more physicians (at least one oncologist and one BMT physician).
  * Arm E: Neuroblastoma ** Neuroblastoma (ICD-O morphology 9500/3) or ganglioneuroblastoma (nodular or intermixed) verified by histology or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites.
* Disease Status at Enrollment

  * Arm A, Arm B and Arm D must have fit one of the following:

    * no evidence of disease or
    * stable, non-progressive disease (defined as non-progressive abnormalities on physical exam or CT and/or MRI) within 4 weeks of study entry
  * Arm C: Evidence of progressive or recurrent GCT (measurable or non-measurable) following one or more cisplatin-based chemotherapy, defined as meeting at least one of the following criteria:

    * Tumor biopsy of new or growing or unresectable lesions demonstrating viable non-teratomatous GCT. Patients with incomplete gross resection where viable GCT is found are considered eligible.
    * Consecutive elevated serum tumor markers (HCG or AFP) that are increasing. Increase of an elevated LDH alone does not constitute progressive disease.
    * Development of new or enlarging lesions in the setting of persistently elevated HCG or AFP, even if the HCG and AFP are not continuing to increase.
  * Arm E: Patients with the following disease stages at diagnosis are eligible, if they meet the other specified criteria.

    * Patients with newly diagnosed neuroblastoma with INSS Stage 4 are eligible with the following:

      * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features or
      * Age > 18 months (> 547 days) regardless of biologic features or
      * Age 12-18 months (365-547 days) with any of the following 3 unfavorable biologic features (MYCN amplification, unfavorable pathology and/or DNA index = 1) or any biologic feature that is indeterminate/unsatisfactory/unknown.
    * Patients with newly diagnosed neuroblastoma with INSS Stage 3 are eligible with the following:

      * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features or
      * Age > 18 months (> 547 days) with unfavorable pathology, regardless of MYCN status.
    * Patients with newly diagnosed neuroblastoma with INSS Stage 2A/2B with MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features.
    * Patients with newly diagnosed neuroblastoma with INSS Stage 4S with MYCN amplification (> 4-fold increase in MYCN expression signals as compared to reference signals), regardless of additional biologic features.
    * Patients ≥ 365 days initially diagnosed with neuroblastoma INSS Stage 1, 2, 4S who progressed to aStage 4 without interval chemotherapy.
* Age and Performance Status

  * Age and Performance Status, Arm A

    * Age: 0 - 70 years
    * Performance status: Karnofsky Performance Status ≥ 50% for patients > 16 years of age or Lansky Play Score ≥ 50 for patients ≤ 16 years of age (Note: Neurologic deficits in patients with CNS tumors must be stable for a minimum of 1 week prior to study entry)
  * Age and Performance Status, Arm B

    * Age: see Eligible diseases, section 3.1, for age criteria
    * Performance status: Karnofsky Performance Status ≥ 50% for patients > 16 years of age or Lansky Play Score ≥ 50 for patients ≤ 16 years of age (Note: Neurologic deficits in patients with CNS tumors must be stable for a minimum of 1 week prior to study entry)
  * Age and Performance Status, Arm C

    * Age: 0-70 years of age
    * Performance status: Karnofsky Performance Status ≥ 70% for patients > 16 years of age or Lansky Play Score ≥ 70 for patients ≤ 16 years of age
  * Age and Performance Status, Arm D

    * Age: see Eligible diseases, section 3.1, for age criteria
    * Performance status: Karnofsky Performance Status ≥ 50% for patients > 16 years of age or Lansky Play Score ≥ 50 for patients ≤ 16 years of age (Neurologic deficits in patients with CNS tumors must be stable for a minimum of 1 week prior to study entry)
  * Age and Performance Status, Arm E

    * Age: Patients must be ≤ 30 years of age at the time of initial diagnosis.
    * Performance status: Karnofsky Performance Status ≥ 50% for patients > 16 years of age or Lansky Play Score ≥ 50 for patients ≤ 16 years of age
* Organ Function

  * Organ Function, Arm A

    * Hematologic: hemoglobin of >9 gm/dl and platelet count > 20,000/μl. Patients may receive transfusions as necessary.
    * Renal: GFR ≥ 50 ml/min/1.73m2 or serum creatinine ≤ 2.5 x ULN for age
    * Hepatic: AST or ALT ≤ 5 x ULN and bilirubin ≤ 5 x ULN
    * Cardiac: ejection fraction ≥ 45% or no clinical evidence of heart failure
    * Pulmonary: oxygen saturation > 92% at rest (on room air)
  * Organ Function, Arm B (to begin first consolidation cycle)

    * Timing: patients must be fully recovered from radiation, induction chemotherapy or surgery prior to receiving consolidation, with minimum elapsed time of 2 weeks.
    * Hematologic: ANC > 750/μl, hemoglobin of >8 gm/dl (may receive PRBC transfusions) and platelet count > 75,000/μl (transfusion independent).
    * Renal: GFR ≥ 50 ml/min/1.73m2
    * Hepatic: AST or ALT ≤ 2.5 x ULN and bilirubin ≤ 1.5 x ULN
    * Cardiac: ejection fraction ≥ 45% or no clinical evidence of heart failure
    * Pulmonary: oxygen saturation > 94% at rest (on room air)
    * Central Nervous System: patients with seizure history are allowed if on anti-convulsants and well controlled; patients must not be in status epilepticus, coma or require assisted ventilation
  * Organ Function, Arm C (to begin TI chemotherapy)

    * Hematologic: ANC ≥ 750/mm3, platelets ≥ 75,000/mm3
    * Renal: GFR ≥ 50 ml/min/1.73m2 or serum creatinine ≤ 2.5 x ULN for age
    * Hepatic: AST or ALT ≤ 2.5 x upper limits of normal (ULN), if hepatic involvement < 5 x ULN; bilirubin ≤ 2.0 x upper limits of normal (ULN)
  * Arms A and C: Patients with a history of CNS tumor involvement are eligible if they have completed treatment for CNS disease (radiotherapy or surgery or chemotherapy), have recovered from or stabilization of the side effects associated with the therapy and have no evidence of progressive CNS disease at the time of enrollment
  * Organ Function, Arm D

    * Timing: patients must be fully recovered from radiation, induction chemotherapy or surgery prior to receiving consolidation, with minimum elapsed time of 2 weeks.
    * Hematologic: ANC > 750/μl, hemoglobin of >8 gm/dl (may receive PRBC transfusions) and platelet count > 75,000/μl (transfusion independent).
    * Renal: GFR ≥ 50 ml/min/1.73m2
    * Hepatic: AST or ALT ≤ 2.5 x ULN and bilirubin ≤ 1.5 x ULN
    * Cardiac: ejection fraction ≥ 45% or no clinical evidence of heart failure
    * Pulmonary: oxygen saturation > 92% at rest (on room air)
    * Central Nervous System: patients with seizure history are allowed if on anti-convulsants and well controlled; patients must not be in status epilepticus, coma or require assisted ventilation
  * Organ Function, Arm E

    * No evidence of disease progression: defined as increase in tumor size of >25% or new lesions.
    * Timing: Recovery from last induction course of chemotherapy.
    * Minimum frozen PBSC of 4 x 106 CD34 cells/kg as 2 aliquots; i.e. 2 x 106 CD34 cells/kg for each transplant are mandatory. A third aliquot of 2 x 106 CD34 cells/kg is strongly recommended for back-up.
    * Hepatic: AST < 3 x upper normal
    * Cardiac: Shortening fraction ≥ 27%, or ejection fraction ≥ 50%, no clinical congestive heart failure.
    * Renal: Creatinine clearance or GFR > 60 ml/min/1.73m2 (If a creatinine clearance is performed at end of induction and the result is < 100 ml/min/1.73m2, a GFR must be performed using a nuclear blood sampling method or iothalamate clearance method. Camera method is NOT allowed as measure of GFR prior to or during Consolidation therapy for patients with GFR or creatinine clearance of < 100 ml/min/1.73m2.)

Exclusion Criteria:

* Arm A, B, C, and D:

  * Pregnant or breastfeeding
  * Active, uncontrolled infection and/or human immunodeficiency virus (HIV) positive constitute progressive disease.
  * Concomitant enrollment on clinical study (such as COG study) that does not allow co-enrollment on this standard of care protocol (Arm B only)
* Arm E: Pregnant or breastfeeding

  * Active, uncontrolled infection and/or HIV positive
  * Known contraindication to PBSC collection. Examples of contraindications might be a weight or size less than that determined to be feasible at the collecting institution, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure.
  * Patients that are 12-18 months of age with INSS Stage 4 and all 3 favorable biologic features (ie, non- amplified MYCN, favorable pathology, and DNA index > 1).

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 Year
  Number of patients who have received autologous transplant for high risk or relapsed solid tumor and certain CNS tumors and are alive at 1 year.

SECONDARY OUTCOMES:
Number of Patients Who Achieved Transplant Engraftment | Day 42
  Engraftment is defined as absolute neutrophil recovery > 500 cells/ul.
Disease Free Survival | 1 Year
  Number of patients who do not have evidence of disease returning after transplant (alive and in remission).
Treatment-Related Mortality | Day 100
  Number of patients died due to treatment received.
Disease Free Survival | 3 Years
  Number of patients who do not have evidence of disease returning after transplant (alive and in remission).

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Gupta, MBBS, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States